CLINICAL TRIAL: NCT06549478
Title: A Pilot Study of BgRT for Bone Metastases
Brief Title: Biology-Guided Radiation Therapy for the Treatment of Patients With Bone Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23937; NCI-2024-06473 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23937 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy, Image-Guided; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (BgRT) (Experimental): Patients undergo a single fraction of BgRT on day 0. Patients undergo PET/CT on study and optionally during follow up.
  Interventions: Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Radiation: Image Guided Radiation Therapy — Undergo BgRT
  Other Names: IGRT; image-guided radiation therapy; Image-Guided Radiotherapy
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests the safety and effectiveness of a single-dose treatment of biology-guided radiation therapy (BgRT) in treating patients with painful cancer that has spread from where it first started (primary site) to the bone (bone metastases). Bone metastases can result in significant pain and reduction in quality of life. Single fraction radiation therapy (SFRT) can produce equivalent pain relief compared to multi-fraction radiation therapy, but SFRT treatments generally lead to higher rates of retreatment. BgRT is a new and innovative form of radiation delivery that uses a signal generated by positron emission tomography to guide external beam radiation therapy. It is a technology breakthrough that uses live, continuously updated data throughout the entire treatment session to determine exactly where to deliver radiotherapy to biologically active tumors. Giving BgRT may be safe and effective in treating patients with painful bone metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate pain response by 14 gray (Gy) single fraction (SF)-BgRT for patients with painful bone metastases.

SECONDARY OBJECTIVE:

I. To evaluate patient-reported health related quality of life (QOL), clinician-rated toxicity per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0, radiographic evidence of disease progression at treated sites, and rate of re-irradiation.

OUTLINE:

Patients undergo a single fraction of BgRT on day 0. Patients undergo positron emission tomography (PET)/computed tomography (CT) on study and optionally during follow up.

After completion of study treatment, patients are followed up at 2 weeks, 3 months and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Pathologic diagnosis of cancer
* Painful bone metastases from any solid cancers (i.e., a score of at least 2 on a 0-10 scale, 0 representing no pain and 10 representing maximum pain)
* Concurrent treatment of up to 3 radiation fields is allowed
* Standardized uptake value maximum (SUVmax) of the target bone lesions on diagnostic PET > 6
* Size of the target bone lesion 1.5-5 cm
* Pre-screening assessment confirms that the intervention can be administered without exceeding dose constraint guidelines
* Patients with brain metastases can be included but brain metastases must be treated prior to enrollment and follow up magnetic resonance imaging (MRI) 3 months after treatment shows stable findings
* Life expectancy ≥ 6 months in the opinion of the treating investigators
* Off systemic therapy for at least one week prior and one week after study intervention
* Patients able to complete pain assessment and quality of life surveys who do not have cognitive impairment

Exclusion Criteria:

* Patients with prior radiation therapy to the treatment sites
* Untreated spinal cord compression
* Pathologic fracture at the evaluated site
* Serious medical comorbidities precluding radiotherapy
* Unable to undergo a PET/CT scan
* Pregnant and/or breastfeeding women are excluded from this study as these agents may have the potential for teratogenic or abortifacient effects
* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics, patients who exhibit cognitive impairments/ who are unable to complete study materials: assessments/questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year follow-up
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Toxicity is defined as any ≥ grade 3 gastrointestinal, genitourinary, lung, or skeletomuscular toxicities that is considered at least possibly related to the study treatment and occurs within 3 months after the treatment.
Pain response | Up to 1 year follow-up
  Will be assessed using international consensus endpoints assessing a combination of pain severity and analgesic consumption. Pain progression reflects either (a) an increase in a worst-pain score of 2 or more without reduced daily morphine milligram equivalent (MME), or (b) no change in worst-pain score or 1 point above baseline and an increase in daily MME of at least 25%. Indeterminate response then indicates all other responses. Overall response is defined as sum of complete response and partial response at 3 months after single fraction-biology-guided radiation therapy.

SECONDARY OUTCOMES:
Rates of re-irradiation | At 1 year follow-up
Radiographic evidence of disease progression | Up to 1 year follow-up
  Radiographic evidence of disease progression at treated sites will be assessed using imaging scans.
Patient-reported health related quality of life (QOL) | Up to 1 year follow-up
  QOL will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Bone Metastases Module.
Incidence of clinician-related chronic toxic effects | Up to 1 year follow-up
  Toxicity is defined as any ≥ grade 3 gastrointestinal, genitourinary, lung, or skeletomuscular toxicities that is considered at least possibly related to the study treatment and occurs within 3 months after the treatment. Clinician-related chronic toxic effects will be assessed using the Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States